CLINICAL TRIAL: NCT00537030
Title: Pharmacology and Toxicity of Erwinia Asparaginase (Erwinase?; Crisantaspase; IND 290) Following Allergy to PEG-Asparaginase in Treatment of Children With Acute Lymphoblastic Leukemia (ALL)
Brief Title: Erwinia Asparaginase After Allergy to PEG-Asparaginase in Treating Young Patients With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AALL07P2; NCI-2009-00316 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 07-162; COG-AALL07P2; CDR0000566349; AALL07P2 (Other: Childrens Oncology Group); AALL07P2 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Adult Acute Lymphoblastic Leukemia; Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; Leyk

ARMS (1):
- Treatment (chemotherapy) (Experimental): Patients receive 6 doses of Erwinia asparaginase IM on a Monday/Wednesday/Friday schedule as a replacement for each scheduled dose of PEG-asparaginase remaining on the original treatment protocol. All other chemotherapy continues according to the original treatment protocol.
  Interventions: Drug: Asparaginase; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Asparaginase — Given IM
  Other Names: ASP-1; Asparaginase II; Asparaginase-E.Coli; Colaspase; Elspar; Kidrolase; L-Asnase; L-ASP; L-Asparaginase; L-Asparagine amidohydrolase; Laspar; Lcf-ASP; Leucogen; Leunase; MK-965; Paronal; Re-82-TAD-15; Serasa; Spectrila
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This clinical trial is studying the side effects of Erwinia asparaginase and what happens to the drug in the body in treating young patients with acute lymphoblastic leukemia who are allergic to PEG-asparaginase. Drugs used in chemotherapy, such as Erwinia asparaginase, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the 48-hour trough serum asparaginase activity is ? 0.1 IU/mL in young patients with acute lymphoblastic leukemia treated with Erwinia asparaginase after allergy to PEG-asparaginase.

II. To determine the frequency of asparaginase-related toxicity in these patients.

III. To characterize the pharmacokinetics of Erwinia asparaginase in these patients.

SECONDARY OBJECTIVES:

I. To compare serum asparaginase activity and serum asparagine concentration between patients treated with Erwinia asparaginase on this trial and historical controls treated with PEG-asparaginase on CCG-1961 and CCG-1962.

II. To determine the 72-hour serum asparaginase activity on days 8 or 11 or 13 based on the starting date of Erwinia asparaginase therapy.

III. To determine the presence of anti-Erwinia asparaginase antibodies in patients treated with a course(s) of Erwinia asparaginase following clinical allergy to PEG-asparaginase (PEG, pegaspargase).

IV. To determine if serum asparagine is adequately depleted on days 12 or 13 in a subset of these patients.

OUTLINE: This is a multicenter study.

Patients receive 6 doses of Erwinia asparaginase intramuscularly (IM) on a Monday/Wednesday/Friday schedule as a replacement for each scheduled dose of PEG-asparaginase remaining on the original treatment protocol. All other chemotherapy continues according to the original treatment protocol.

Blood samples are collected periodically for pharmacokinetic, pharmacodynamic, and antibody studies.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia
* Concurrently enrolled on a frontline Children's Oncology Group treatment trial (i.e., COG-AALL0232 or COG-AALL0531, COG-AALL0331, or COG-AALL0434) at a participating institution

  * Must have 1 or more courses of asparaginase remaining to be administered on the treatment protocol
* Must have had a grade ? 2 hypersensitivity reaction to PEG-asparaginase
* No history of pancreatitis ? grade 2
* No prior Erwinia asparaginase

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2008-02-11 (Actual); Primary Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Salzer, Principal Investigator — Children's Oncology Group
Locations (43):
- United States (43):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Confirmation of the patient ineligibility was not confirmed by the COG study team until the patient received their first dose of Erwinia. Patient was removed from the COG frontline study (AALL08P1) prior to enrollment of this study.
Groups:
- Erwinia Asparaginase: Patients receive 6 doses of Erwinia asparaginase (dosage 25,000 IU/m2 intramuscularly (IM) on a Monday/Wednesday/Friday schedule as a replacement for each scheduled dose of PEG-asparaginase remaining on the original treatment protocol. All other chemotherapy continues according to the original treatment protocol.
  pharmacological study : Correlative studies
  laboratory biomarker analysis : Correlative studies
  asparaginase : Given IM
Period: Overall Study
Arm/Group | Erwinia Asparaginase
Started | 59
Completed | 43
Not Completed | 16
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 2
Not completed — ≥ Grade 2 allergy | 7
Not completed — Disease progression/ relapse during Tx | 1
Not completed — Ineligible | 2
Not completed — Inevaluable | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erwinia Asparaginase
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 46
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Trough Serum Asparaginase Activity ≥ 0.1 IU/mL
Description: Percentage of participants who had trough serum asparaginase activity ≥ 0.1 IU/mL in the blood 48 hours post administration of Erwinia asparaginase
Time Frame: 48 hours post administration of Erwinia asparaginase
Population: Of the 59 enrolled participants, there were 2 ineligible and 2 in-evaluable participants. From the remaining 55 participants, 52 participants had an acceptable sample that could be reported on.
Measure: Number; unit: Percent of participants
Arm/Group | Erwinia Asparaginase
Number analyzed (Participants) | 52
Percent of participants | 94.5

2. Secondary Outcome: Determine if Plasma Asparagine is Adequately Depleted
Description: Plasma asparagine depletion will be determined in a subset of 20 patients limited to participating Phase I Institutions.
Time Frame: On days 12 or 13
Population: No data available for this analysis.
Arm/Group | Erwinia Asparaginase
Number analyzed (Participants) | 0

3. Secondary Outcome: Presence of Anti-Erwinia Asparaginase Antibodies in Children Treated With a Course(s) of Erwinase® Following Clinical Allergy to PEG-asparaginase
Description: An ELISA (enzyme-linked immunosorbent assay) method will be used to determine the presence of specific anti-Erwinia and anti-PEG-asparaginase antibodies at baseline, and of specific anti-Erwinia asparaginase antibodies after first and subsequent exposures to Erwinase®. The rate of antibody formation will be described and compared informally to experience in CCG-1962 and 1961. Serum asparaginase activity will be compared during Erwinase® courses as an indication of the neutralizing effect of antibodies on the enzyme effect.
Time Frame: At baseline, prior to doses 4, 5, and 6 and on days 15 and 22
Population: no data available for this analysis.
Arm/Group | Erwinia Asparaginase
Number analyzed (Participants) | 0

4. Secondary Outcome: Percentage of Participants Who Experienced Toxicities
Description: The percentage of participants who experienced toxicities: Allergy rate, Hyperglycemia Rate, Pancreatitis Rate, Hemorrhage/Thrombosis Rate
Time Frame: up to 1 year
Population: Patients who had toxicity data collected.
Measure: Number; unit: percentage of participants
Arm/Group | Erwinia Asparaginase
Number analyzed (Participants) | 55
percentage of participants
  Allergy Rate | 10.9
  Hyperglycemia Rate | 10.9
  Pancreatitis Rate | 1.8
  Hemorrhage/Thrombosis Rate | 0

ADVERSE EVENTS:
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution, via expedited reporting (NCI AdEERs / CAeRs). The "AE Other" table reflects all CTCAEs collected excluding those that were reported as SAEs. There were 2 ineligible and 2 in-evaluable patients excluded from reporting of adverse events, leaving a total of 55 participants included in the AE
Arm/Group | Erwinia Asparaginase
Serious Adverse Events (participants affected / at risk) | 9/55
Other Adverse Events (participants affected / at risk) | 15/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erwinia Asparaginase (N=55)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Allergic reaction (Immune system disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 3
Blood bilirubin increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erwinia Asparaginase (N=55)
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 1
Allergic reaction (Immune system disorders) | 4
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 4
Lipase increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No